CLINICAL TRIAL: NCT05198531
Title: Phase Ib Clinical Study to Evaluate the Safety and Efficacy of TQB2858 Injection to the Subjects With Recurrent/Metastatic Nasopharyngeal Cancer
Brief Title: To Evaluate the Safety and Efficacy of TQB2858 Injection to the Subjects With Recurrent/Metastatic Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-Ib-01
Record Dates: First submitted 2022-01-19; First posted 2022-01-20 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Recurrent / Metastatic Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 Injection combining with other drugs (Experimental): Combination 1 is TQB2858 Injection and Anlotinib Hydrochloride Capsules. Combination 2 is TQB2858 Injection, Gemcitabine Hydrochloride Injection and Cisplatin Injection for 4-6 cycles of induction chemotherapy, then using TQB2858 Injection and Anlotinib Hydrochloride Capsules for maintenance treatment.
  Combination 3 is TQB2858 Injection, Gemcitabine Hydrochloride Injection, Cisplatin Injection and Anlotinib Hydrochloride Capsules for 4-6 cycles of induction chemotherapy, then using TQB2858 Injection and Anlotinib Hydrochloride Capsules for maintenance treatment.
  Interventions: Drug: TQB2858 Injection; Drug: Anlotinib Hydrochloride Capsule; Drug: Gemcitabine hydrochloride injection; Drug: Cisplatin Injection

INTERVENTIONS:
Drug: TQB2858 Injection — TQB2858 Injection, a bifunctional fusion protein against Programmed death ligand 1 (PD-LI) and transforming growth factor-β (TGF-β). TQB2858 Injection blocks the PD-1/PD-L1 pathway and neutralizes TGF-β in the tumor microenvironment.
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
Drug: Gemcitabine hydrochloride injection — Gemcitabine hydrochloride, cell cycle-specific antimetabolites, mainly acting on tumor cells in the DNA synthesis phase (S phase cell). Under certain conditions, it can prevent the progression from G1 phase to S phase.
Drug: Cisplatin Injection — After cisplatin enters cells, it reacts with DNA to form cross-links between two points or two strands in DNA, thereby inhibiting DNA replication and transcription, resulting in DNA breaks and miscoding.

SUMMARY:
This study is a single-arm, randomized, open-label, multi-cohort Phase Ib clinical trial. The experimental drug is TQB2858 Injection. The trial was divided into 3 cohorts. Cohort 1 included patients with advanced nasopharyngeal carcinoma who had previously failed platinum-based chemotherapy and immune checkpoint inhibitors (programmed cell death protein 1 (PD-1)/ Programmed death-ligand 1 (PD-L1), etc.). Cohorts 2 and 3 were randomized into patients with advanced, untreated nasopharyngeal carcinoma who had not received prior systemic therapy. A total of 60-90 subjects are required.

ELIGIBILITY:
Inclusion Criteria:

* 1 Voluntarily joined the study and provide written informed consent and authorization permitting release of Protected Health Information.
* 2 Male or female patient ≥18 and ≤75 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥12 weeks.
* 3 Histologically or cytologically proven diagnosis of nasopharyngeal cancer (NPC), Stage IVb or not amenable for or local treatment (based on 2017, the 8th edition of the American Joint Committee on Cancer (AJCC) staging system of tumor-node-metastasis (TNM) of nasopharyngeal cancer).
* 4 Subject meets one of the following criteria:

  * Arm 1: Progression (Tumor-imaging proven) after platinum-based chemotherapy and Tumor Immunotherapy (PD-1/PD-L1 Checkpoint Inhibitors, etc.).
  * Attention: Progression during therapy or after therapy within 6 months, neoadjuvant/ adjuvant therapy, radical chemoradiotherapy are considered as the first-line treatment.
  * Arm 2 and 3: Not received systemic anti-tumor therapy for recurrent / metastatic nasopharyngeal cancer.
  * Attention: Progression after therapy more than 6 months, neoadjuvant/ adjuvant therapy, radical chemoradiotherapy are not considered as the first-line treatment.
* 5 Have at least 1 measurable disease defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
* 6 Have adequate baseline function and performance status：

  * a) Standard hematology test (no blood or product transfusions for a period of at least 7 days prior to enrollment).

    i. Hemoglobin (HGB) >90 g/L; ii. Neutrophil count (NEUT) ≥1.5 × 109/L; iii. Platelets (PLT) ≥75 × 109/L;
  * b) Serum chemistry i. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 upper limit of normal (ULN) or ≤ 5 x ULN for subjects with hepatic metastatic tumor; ii. Bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN for subjects with Gilbert Syndrome; iii. Creatinine ≤ 1.5 x ULN or Creatinine Clearance ≥ 60 mL/min;
  * c) Blood Coagulation Test i. Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR) and Prothrombin Time (PT) ≤ 1.5 (No anticoagulant therapy);
  * d) left ventricular ejection fraction (LVEF) ≥ 50%;
* 7 Women of child-bearing potential must agree to use contraceptive method(s) throughout the study and for at least 180 days after the last dose of assigned treatment. Serum pregnancy test negative within 7 days before enrollment and must be non-lactating.

Exclusion Criteria:

* 1 Complicated disease and history:

  1. Has developed other malignant tumors within 3 years or is currently suffering from;
  2. With factors affecting take medicine orally (such as unable to swallow drugs or bowel obstruction, etc.)
  3. Unmitigated toxic reactions above Common Terminology Criteria for Adverse Events (CTCAE) grade 1 due to any prior treatment, excluding hair loss and peripheral sensory nerve disorders related to platinum-based chemotherapy;
  4. Received major surgical treatment, significant traumatic injury or long-term unhealed wounds or fractures (excluding needle biopsy for diagnosis, endoscope, etc.) within 28 days prior to the commencement of study treatment;
  5. With arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage), deep venous thrombosis and pulmonary embolism;
  6. With active pulmonary tuberculosis, idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment or active pneumonia with clinical symptoms;
  7. History of psychotropic substance abuse and inability to quit or with mental disorders;
  8. Received allogeneic bone marrow transplantation or solid organ transplantation;
  9. Subjects with any severe and/or uncontrolled disease:

     * i. Uncontrolled hypertension (defined as systolic BP >150 mm Hg or diastolic BP > 100 mm Hg pressure)
     * ii. Grade 2 or greater cardiac ischemia, myocardial infarction or cardiac arrhythmia (including QTc ≥ 480 ms) ;and New York Heart Association (NYHA) Grade II or greater congestive heart failure;
     * iii. Active or uncontrolled infections;
     * iv. Decompensated liver cirrhosis and active hepatitis (Hepatitis B reference: HBsAg positive, and HBV DNA> 2500 copy/mL or > 500 IU/mL; Hepatitis C reference: HCV antibody positive, and HCV RNA > ULN);
     * v. Renal failure requiring hemodialysis or peritoneal dialysis；
     * vi. Known history of immunodeficiency infection;
     * vii. Urinalysis：urine protein ≥ ++，and confirmed 24-hour urinary protein > 1.0g;
* 2 Tumor-related symptoms and treatment:

  1. History of surgery, chemotherapy, radiation or other anti-tumor therapy within 4 weeks prior to enrollment (calculated from the date of the last dose);
  2. History of Chinese patent drugs with anti-tumor indications approved by National Medical Products Administration (NMPA) (including compound cantharide capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea oil injection/capsule, Xiaoaoping tablet/injection, Huabenin capsule, etc.) within 2 weeks before enrollment;
  3. History of Tumor Immunotherapy of TGF-β inhibition;
  4. Previously received bevacizumab, arotinib, apatinib, renvatinib or other anti-vascular targeted drug therapy;
  5. History of secondary radiotherapy;
  6. Imaging (CT or MRI) evidence of tumor invading the significant blood vessels or likely to invade and cause fatal massive bleeding during study, accessed by investigators;
  7. With uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
  8. Known uncontrolled or symptomatic active central nervous system (CNS) metastasis (characterized by clinical symptoms, brain edema, spinal cord compression, cancerous meningitis, leptomeningeal disease and /or progressive growth); (exclude those, with the history of CNS metastasis or spinal cord compression, clinical symptoms stabilized less than 4 weeks after discontinuation of dehydrants and steroids);
* 2 Research Treatment Related:

  1. History of live attenuated vaccine vaccination within 28 days prior to enrollment or planing of live attenuated vaccine vaccination during the study period;
  2. Definite bleeding tendency or bleeding symptoms with significant clinical significance within 28 days prior enrollment, including gastrointestinal bleeding, nasal bleeding (excluding epistaxis and retractive runny nose), and with hemorrhagic diseases or coagulation disorders;
  3. History of hemoptysis or hemoptysis within 28 days prior enrollment (defined as coughing or coughing out ≥ 1 teaspoon of blood or small blood clots or only coughing up blood without sputum) , blood in sputum are not excluded;
  4. Severe allergy history of antibody drugs or others;
  5. History of active autoimmune disease requiring systemic treatment within 2 years prior to enrollment (e.g. palliative drugs, corticosteroids, or immunosuppressants) .

     * i. Including autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism or multiple sclerosis;
     * ii. Exclude Skin diseases without systemic treatment, such as vitiligo, psoriasis and hair loss；
     * iii. Including asthma requiring medical intervention with bronchodilators;
     * iv.Alternative therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered as systemic therapy;
  6. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. (dose of >10mg/ day prednisone or other equivalent efficacy hormone), and continued to use within 2 weeks prior to enrollment;
* 4 History of participating in other anti-tumor clinical trials in the previous 4 weeks;
* 5 Other damage to the safety of patients or other situations affecting patients to complete the study, assessed by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | Baseline up to PD/die, about 20 months
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | Baseline to CR/PR, about 16 months
  The percentage of participants with a best overall response defined as complete response (CR) or partial response (PR).
Progression-free survival (PFS) | Baseline to PD/die, about 20 months
  The time from enrollment to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
Disease Control rate (DCR) | Baseline to CR/PR/SD, about 16 months
  Calculated as the percentage of participants with best overall response of CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD).
Duration of Overall Response (DOR) | Baseline up to PD/die, about 20 months
  The time from the date of participants with a first overall response defined as complete response (CR) or partial response (PR) to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
Overall survival (OS) | Baseline up to die, about 46 months
  The time from enrollment to the time of death from any cause.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - Guangxi Tumor Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Hunan Cancer Hospital, Changsha, Hunan